CLINICAL TRIAL: NCT03267654
Title: Gefitinib Versus Combination of Gefitinib With Chemotherapy or Anti-angiogenesis as 1st Line Treatment in Advanced NSCLC Patients Detected With Bim Deletion or Low EGFR Activating Mutation Abundance：A Randomized, Multicentre, Phase II Study
Brief Title: Gefitinib With Chemotherapy or Anti-angiogenesis in NSCLC Patients With Bim Deletion or Low EGFR Mutation Abundance
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Qilu Pharmaceutical Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: SHENKANG
Record Dates: First submitted 2017-08-14; First posted 2017-08-30 (Actual); Last update posted 2020-08-03 (Actual); Status verified 2020-07

CONDITIONS: Non-small-cell Lung Cancer
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung | interventions — Drug Therapy; apatinib

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- gefitinib combined with chemotherapy (Experimental): gefitinib 250mg Qd combined with pemetrexed plus carboplatin: pemetrexed (500mg/m²day 1 intravenously) plus carboplatin (AUC=5,day 1,intravenously) every 21 days.
  Interventions: Drug: gefitinib combined with chemotherapy
- gefitinib combined with apatinib (Experimental): gefitinib 250mg Qd combined with apatinib 250mg per 21 days
  Interventions: Drug: gefitinib combined with apatinib
- gefitinib single agent (Active Comparator): Advanced NSCLC patients with EGFR activating mutation (L858R, 19Del) received gefitinib 250mg Qd orally until progression, intolerable toxicity or death.
  Interventions: Drug: gefitinib single agent

INTERVENTIONS:
Drug: gefitinib combined with chemotherapy — Gefitinib 250mg, p.o., q.d., continuous regimens on an empty stomach or after meal for 2 hours until disease progression, intolerable toxicity or patient withdraw ICF.
  Pemetrexed (500mg/m²day 1 intravenously) plus carboplatin (AUC=5,day 1,intravenously) every 21 days. Every 3 weeks is a chemotherapy cycle, and 4 chemotherapy cycles is maximum limit.
  Other Names: yiruike
  Arms: gefitinib combined with chemotherapy
Drug: gefitinib combined with apatinib — gefitinib 250mg, p.o., q.d., continuous regimens on an empty stomach or after meal for 2 hours.
  Apatinib 250mg, p.o., q.d. per 21 days. until disease progression, intolerable toxicity, patient withdraw ICF or death.
  Other Names: yiruike
  Arms: gefitinib combined with apatinib
Drug: gefitinib single agent — Patients received Gefitinib 250mg q.d. orally until disease progression, intolerable toxicity or death.
  Other Names: yiruike
  Arms: gefitinib single agent

SUMMARY:
This is an open-label, multicenter, randomized, phase II clinical trial, which aims to evaluate the effectiveness and safety of gefitinib versus combination of gefitinib and doublet chemotherapy or apatinib in advanced non-small cell lung cancer (NSCLC) patients with epidermal growth factor receptor (EGFR) activating mutation (exon 19 deletion or exon 21 L858R point mutation), accompanied with Bim deletion or low activating EGFR mutation abundance.

DETAILED DESCRIPTION:
BIM (bcl-2 interacting mediator of cell death) deletion polymorphism and low EGFR mutation abundance were poor clinical response markers to epidermal growth factor receptor tyrosine kinase inhibitors (EGFR-TKIs) in NSCLC patients who had EGFR mutations.This is a phase II clinical trial to investigate the efficacy of combination treatment for patients harboring above risk factors.

Advanced EGFR mutated NSCLC Patients with Bim deletion or EGFR low mutation abundance were randomized divided into following three treatment groups:

A: gefitinib 250mg Qd combined with doublet chemotherapy: pemetrexed (500mg/m²，day 1 ，intravenously) plus carboplatin (AUC=5,day 1,intravenously) every 21 days.

B: gefitinib 250mg Qd combined with apatinib 250mg/d intravenously per 21 days. C: gefitinib 250mg Qd

ELIGIBILITY:
Inclusion Criteria:

1. Volunteered for attending the study, and signed informed consent form (ICF)to participate in the study.
2. Cytologically and Histologically documented, locally advanced or recurrent or metastatic (stage IIIb, IIIc, IV) non-small cell lung cancer patients .
3. EGFR mutation (exon 19 deletion or exon 21 L858R) with Bim deletion or low abundance for EGFR mutation.
4. Age range: 18 years to 75 years.
5. Patients must have measurable lesion according to the RECIST (version 1.1) criteria.
6. Life expectancy of ≥ 12 weeks
7. ECOG (Eastern Cooperative Oncology Group) performance status of ≤ 1.
8. Patients hadn't received past system treatment, including cytotoxic drugs; For patients who have received adjuvant or neoadjuvant chemotherapy appears recurrence or metastasis more than 6 months from accepting the last dose of chemotherapy drugs
9. Adequate organ function as defined by the following criteria:

   * Bone marrow function: absolute neutrophil count ≥ 1,500,000,000/L and platelet count ≥100,000,000,000/L and hemoglobin ≥9g/dL.
   * Liver function: Total bilirubin ≤ 1.5 ULN (upper limit of normal). AP (alkaline phosphatase), AST ( aspartate aminotransferase) and ALT (alanine transaminase) ≤ 3 ULN in the absence of liver metastases or up to 5 ULN in case of liver metastases.
   * Renal function: creatinine clearance ≥ 60 ml/min. (based on modified Cockcroft-Gault formula).
   * INR （international normalized ratio）≤ 1.5, and partial thromboplastin time (PTT) or activated partial thromboplastin time (aPTT) ≤ 1.5 ULN.
10. For all females of childbearing potential a negative serum/urine pregnancy test must be obtained within 48 hours before enrollment. Postmenopausal women must have been amenorrhoeic for at least 12 months to be considered of non-childbearing potential.
11. Fertile men and women must use effective contraception.

Exclusion Criteria:

1. Histology confirmed for squamous carcinomas, including mixed gland scale cancer, small cell lung cancer.
2. Poor controlled hypertension, it means systolic pressure ≥140 mmHg and/or diastolic pressure ≥90 mmHg after drug therapy.
3. There are imaging evidence of tumor invading or closing to the pulmonary vessels (e.g., pulmonary artery, superior vena cava).
4. Thrombosis in 6 months before enrollment, including pulmonary thrombosis or deep venous thrombosis., or patient had medical evidence or history of thrombosis or bleeding tendency regardless of the severity.
5. Patients with medical history of hemoptysis (defined as about 2.5ml bright blood) 2 weeks before the enrollments.
6. Proteinuria ≥++, or 24h proteinuria ≥1.0g.
7. A uncontrolled clinical infection, activity, including but not limited to acute pneumonia.
8. Patients with known liver disease: the hepatitis B virus (HBV) infection and hepatitis b virus DNA (HBV DNA) ≥ 500 copy number or ≥100 IU/ml; or more; or hepatitis C virus (HCV) infection; or liver cirrhosis, etc.
9. Patients who are at risk of human immunodeficiency virus (HIV) or syphilis infection.
10. Patients who have a difficulty in swallowing or drug absorption.
11. There are diseases of alimentary canal such as active duodenal ulcer, the ulcerous colitis, intestinal obstruction or other conditions which can cause gastrointestinal bleeding or perforation in the investigator's opinion; or patient has a history of intestinal perforation, intestinal fistula.
12. Evaluation of cardiac function: left ventricular ejection fraction < 50% (echocardiography); Moderate or above disorders of mitral valve and tricuspid shut down;, serious/unstable angina or acute myocardial infarction coronary artery bypass surgery in 6 months before enrollment; patients with class 2 and above cardiac dysfunction according to New York heart association (NYHA) classification
13. Stroke and transient ischemic in 12 months before enrollment.
14. severe ulcer in the skin wound, trauma and mucosa or fractures have been not fully healed.
15. Patients received CYP3A4 strong inhibitor and/or inducer in 2 weeks before enrollment; Patients received P-gp and breast cancer resistance protein (BCRP) substrates drug in 2 weeks before enrollment.
16. Patients received other anti-tumor treatment at the same time.
17. Patients exist serious psychological or mental abnormalities, so patient compliance is not sufficient.
18. Poorly controlled serous cavity effusion, including but not limited to malignant pleural effusion, malignant pericardial effusion and malignant peritoneal effusion.
19. Patients have a weight loss (≥10%) within 6 weeks before enrollment.
20. The pregnancy of female patients test is positive or lactation women.
21. Patients haven't been diagnosed other malignant disease, except the basal cell carcinoma and cervical carcinoma.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2017-10-12 (Actual); Primary Completion 2020-10-20 (Estimated); Study Completion 2021-12-30 (Estimated)

PRIMARY OUTCOMES:
Progression free survival | 8 weeks
  From start of anti-cancer therapy until progression or death

SECONDARY OUTCOMES:
overall survival | 36 months
  evaluated in the 36th since treatment begain
objective response rate | 8 weeks
  Evaluated the rate of complete response and partial response in the 8 weeks since treatment began
disease control rate | 8 weeks
  Evaluated the rate of complete response，partial response and stable disease in the 8 weeks since anti-cancer therapy
duration of response | 8 weeks
  interval between the time which complete response or partial response happened and progressive disease or death
safety evaluation | 8 weeks
  Safety observation indexes were listed as following: adverse events and serious adverse events (according to CommonTerminology Criteria Adverse Events Version 4.03), physical exam, vital signs(blood pressure, heart rate, respiratory rate,body temperature), weight variation, laboratory examination(hematology, blood biochemistry, urinalysis and so on), electrocardiograph(ECG),ultrasonic cardiogram(UCG), ect.
compare quality of life | 24 months
  Quality of Life Questionnaire(including QLQ-C30 and QLQ-LC13) evaluated since treatment began.At the end of the trial, the differences between the two indicators were compared with Mixed-effects model repeated measures (MMRM), where the baseline was scored as a covariant and the treatment group as a fixed variable. In addition, the baseline values of the two scores, the value of each visit, and the change value of the baseline were statistically described.

CONTACTS AND LOCATIONS:
Overall Officials: Caicun Zhou, Principal Investigator — Shanghai Pulmonary Hospital, Shanghai, China
Locations (1):
- Shanghai Pulmonary Hospital;, Shanghai, Shanghai Municipality, China